CLINICAL TRIAL: NCT01665833
Title: A Retrospective Analysis Determining the Impact of Coronary Anatomy on Angina Relief in Patients Undergoing Coronary
Brief Title: Impact of Coronary Anatomy on Angina Relief in Patients Undergoing Coronary Revascularization
Status: Completed | Type: Observational
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Subhash Banerjee, MD, North Texas Veterans Healthcare System
Other Study IDs: SYNTAX
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Angina; Status Post PCI; Status Post CABG
Keywords: Angina; SYNTAX; Coronary; PCI; CABG
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
We hypothesize that Coronary Artery Disease (CAD) severity assessed by SYNTAX score is an independent predictor of recurrent or persistent angina following coronary revascularization. The SYNTAX score is a score that suggests the severity of coronary artery disease detected by coronary angiography. Coronary revascularization is a procedure that occurs in two ways, a percutaneous coronary intervention (PCI) and a coronary artery bypass graft (CABG) and is done when there is narrowing and blockage or hardening of the arteries (atherosclerosis) surrounding the heart. Narrowing and blockages reduce blood flow to parts of the heart causing chest pain (known as angina) and sometimes myocardial infarction.

DETAILED DESCRIPTION:
PCI and CABG are two well-established revascularization approaches to treatment of chronic angina caused by coronary atherosclerosis. Nevertheless, 35-42% of patients report recurring or persisting anginal symptoms after coronary revascularization. This can be attributed to many structural and functional causes, prominent amongst which is pre-revascularization angina severity, unrevascularized coronary territory, progression of native or bypass graft atherosclerosis, restenosis (re-narrowing of the vessels) and accompanying adjunctive pharmacotherapy.

The SYNTAX score is an angiographic tool for grading the complexity of coronary disease. It is the sum of points assigned to coronary lesions within one of the 16 segments of the coronary tree. The segments are given a 1,2, or 5 based on the disease presence as defined by the American Heart Association classification. The SYNTAX score has been used to help predict the outcomes of patients undergoing PCI with 3-vessel involvement (e.g. a triple bypass or 3-stent placement PCI). Those patients with the highest scores had the highest risk of a poor outcome with PCI revascularization compared to CABG. Despite these observations, the impact of CAD severity on post-revascularization angina, using the SYNTAX has never been systematically addressed in the current era.

ELIGIBILITY:
Inclusion Criteria:

* Any VA patient who has had an PCI from January 1, 2003 and December 31, 2011 and in the database used in protocol 09-018 (VA-CAP Study).
* Any VA patient who has received or will receive a 1-year follow up.

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We propose all patients between January 1, 2003 and December 31, 2011 who underwent an uncomplicated coronary revascularization with PCI and/or CABG for chronic stable angina within the VA. The data set that includes this information is the same as was used for study 09-018 (VA-CAP Study).
Sampling Method: Non-Probability Sample
Enrollment: 4000000 (Actual)
Dates: Start 2003-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Hazard Rate | 1 year follow ups
  Primary and secondary endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Subhash Banerjee, MD, Principal Investigator — Dallas VA Medical Center; Emmanouil Brilakis, MD,PhD, Principal Investigator — Dallas VA Medical Center

REFERENCES:
- [Result] Serruys PW, Morice MC, Kappetein AP, Colombo A, Holmes DR, Mack MJ, Stahle E, Feldman TE, van den Brand M, Bass EJ, Van Dyck N, Leadley K, Dawkins KD, Mohr FW; SYNTAX Investigators. Percutaneous coronary intervention versus coronary-artery bypass grafting for severe coronary artery disease. N Engl J Med. 2009 Mar 5;360(10):961-72. doi: 10.1056/NEJMoa0804626. Epub 2009 Feb 18. PMID 19228612